CLINICAL TRIAL: NCT05356923
Title: PROline and FapI With Late Gadolinium Enhancement in Myocardial Infarction PROFILE-MI - The FAPI Fibrosis Study
Brief Title: PROFILE-MI - The FAPI Fibrosis Study
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 262477; E202251 (Other: University of Edinburgh)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction; Myocardial Fibrosis
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood draw for all participants with recent or prior established myocardial infarction at each attendance for PET/MR scanning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Age- and sex- matched to participants, those aged 50 or over without known heart disease. n=20
  Interventions: Radiation: 68Gallium FAPI PET/MR scan
- Acute myocardial infarction - multi-timepoint imaging: Those aged 50 or over with recent myocardial infarction who will be imaged using PET/MR at 1,2,4, and 12 weeks post-MI. n=20
  Interventions: Radiation: 68Gallium FAPI PET/MR scan
- Acute or chronic myocardial infarction - single timepoint imaging: Those aged 50 or over with recent (n=20) or prior established (>24 months, n=20) myocardial infarction who will be imaged at a single timepoint (1,2,4, or 12 weeks post-MI for acute, at the time of enrolement to the study for chronic).
  Interventions: Radiation: 68Gallium FAPI PET/MR scan

INTERVENTIONS:
Radiation: 68Gallium FAPI PET/MR scan — 68Gallium FAPI PET/MR scan

SUMMARY:
The investigators here propose to investigate the timing and pattern of myocardial fibrosis activity following acute myocardial infarction using hybrid 68Ga-FAPI positron emission tomography and cardiovascular magnetic resonance. The investigators hypothesise that peak fibrosis activity will occur within 2-4 weeks of acute myocardial infarction and will predict subsequent scar formation and cardiac remodelling. Simultaneously, matrix remodelling and fibrosis activity in aortic and coronary atheroma will be assessed enabling the exploration of the presence of unstable atheroma.

DETAILED DESCRIPTION:
Fibrosis is a fundamental process underlying almost all cardiomyopathic conditions. Established fibrosis can be detected by existing imaging techniques including cardiovascular magnetic resonance. However, these techniques are not specific for fibrosis and do not directly measure fibrosis activity or matrix remodelling. This limits the ability to detect early disease and differentiate active from end-stage phenotypes. Fibroblast activation protein is a key factor in fibrogenesis that is expressed in the myocardium following myocardial infarction and in thin-capped fibroatheroma. Radiolabelled fibroblast activation protein inhibitor (68Ga-FAPI) measures in vivo fibrosis activity and matrix remodelling, as supported by preliminary pilot studies. The timing and pattern of myocardial fibrosis activity following acute myocardial infarction will be investigated using hybrid 68Ga-FAPI positron emission tomography. The investigators hypothesise that peak fibrosis activity will occur within 2-4 weeks of acute myocardial infarction and will predict subsequent scar formation and cardiac remodelling. Simultaneously, matrix remodelling and fibrosis activity in aortic and coronary atheroma will also be assessed allowing exploration of the presence of unstable atheroma. This project will enhance understanding of fibrosis activity and matrix remodelling in myocardial infarction and unstable atherosclerotic plaque with potential future application to a broad range of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* specific to cohort;
* aged 50 years or older

Exclusion Criteria:

* Claustrophobia
* Inability to undergo MRI
* eGFR <30ml/min/1.73^m2

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer participants (cohort 1, n=20): those without significant or serious comordibity or known cardiac disease
  Participants with acute myocardial infarction (cohorts 2 and 3, n=40): ST-elevation myocardial infarction within 3 weeks of enrollment
  Participants with chronic myocardial infarction (n=20): ST-elevation myocardial infarction 24 months or more prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Time of maximal fibrosis activity following myocardial infarction | 12 weeks
  SUVmax and TBR of 68Ga-FAPI uptake within the infarct, border zone, and remote myocardium
Whether fibrosis activity predicts myocardial scar volume and ventricular remodelling | 12 months
  As measured by CMR 12 months following acute MI
Fibrosis activity and myocardial remodelling within atherosclerotic plaque in patients with myocardial infarct | 12 weeks
  SUVmax and TBR of 68Ga-FAPI uptake within areas of atherosclerotic plaque in the aorta and/or carotid arteries

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, City Of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barton AK, Craig NJ, Loganath K, Joshi S, Tsampasian V, Mahendran M, Lenell J, Tzolos E, Singh T, Whittington B, Nash J, Williams MC, van Beek EJR, MacAskill MG, Berkeley B, Vezaides S, Brittan M, Baker AH, Sellers S, Fletcher A, Clark T, Waight C, Slart RHJA, Berman D, Dey D, Slomka P, Newby DE, Dweck MR. Myocardial Fibroblast Activation After Acute Myocardial Infarction: A Positron Emission Tomography and Magnetic Resonance Study. J Am Coll Cardiol. 2025 Feb 18;85(6):578-591. doi: 10.1016/j.jacc.2024.10.103. Epub 2025 Jan 8. PMID 39772364